CLINICAL TRIAL: NCT06462768
Title: Neutrophil Extracellular Traps in Systemic Sclerosis
Brief Title: Neutrophil Extracellular Traps in Different Forms of Systemic Sclerosis
Acronym: NETOSE
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO23126
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Systemic Sclerosis; Other Connective Tissue Disease; Systemic Lupus Erythematosus; Dermatomyositis; ANCA Associated Vasculitis
Keywords: Systemic sclerosis; NETosis; polymorphonuclear neutrophil
MeSH Terms: conditions — Scleroderma, Systemic; Lupus Erythematosus, Systemic; Dermatomyositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult with SSc: Adult with SSc
  Interventions: Other: Blood sample
- Other connective tissue disease: Adult with other connective tissue disease
  Interventions: Other: Blood sample
- Control: Healthy adult volunteer
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample to quantify and qualify NETosis in vivo and ex vivo after different stimulations.

SUMMARY:
Systemic SClerosis (SSC) is a systemic disease characterized by limited or diffuse cutaneous sclerosis, microangiopathy, overproduction of autoantibodies and variable organ damage due to vasculopathy and/or fibrosis. The loss of self-tolerance is believed to be caused by the dysregulation of both innate and adaptive immune systems and may involve Reactive Oxygen Species (ROS).

Neutrophils are potent producers of ROS and may play a role in endothelial cells and fibrobasts dysfunction, as in autoantibodies generation. However, their role in SSC pathogenesis remains to be determined. Recent studies discovered abnormal regulation of Neutrophil Extracellular Traps (NETs) in other auto-immune diseases such as Systemic Lupus Erythematosus (SLE). NETs are web-like structures composed of chromatin backbones and granular molecules. They are released by activated neutrophils through a process called "NETosis". Nets were first described in 2004 as a novel host defense mechanism to trap and kill foreign pathogens. Recent evidence shows that NETs also participate in the pathogenesis of a variety of inflammatory and autoimmune diseases, including SLE.

The investigators recently highlighted this phenomenon in SSc, especially in patients with vascular complications and/or at a early stage of the disease. The investigators will now explore the factors implicated in this dysregulation of NETosis in SSc.

DETAILED DESCRIPTION:
This study is designed to assess the role of Neutrophil Extracellular Traps (NETs) in Systemic SClerosis (SSC) as well as to evaluate the correlation between NETs production and NETs composition and the different complications and phenotypes observed in SSC.

100 SSC patients, 30 other connective tissue disease patients and 130 healthy subjects will be recruited. Blood samples will be collected to obtain plasma, serum and polynuclear neutrophils by negative selection.

ELIGIBILITY:
Inclusion Criteria:

*For patients of group 1:

* Patients with systemic sclerosis (ACR-EULAR Criteria)
* Patients taking care of in internal medicine or in dermatology department's of the university hospital of Reims
* Patients consenting to participate to the study
* Patients enrolled in the national healthcare insurance program

For patients of group 2:

* Patients with other connective tissue disease (ACR specific-disease criteria)
* Patients taking care of in internal medicine or in dermatology department's of the university hospital of Reims
* Patients consenting to participate to the study
* Patients enrolled in the national healthcare insurance program

For patients of group 3 (healthy volunteers)

* Patients eligible for blood donation (blood donation regulation criteria of January 11th 2022 decree)
* Patients without medical history of autoimmune systemic or chronic inflammatory systemic disease,
* Patients without current or past neoplasy disease,
* Patients without chronic metabolic pathology
* Patients without treatment by anti inflammatory or corticotherapy for the last 15 days,
* Patients without infectious pathology or inflammatory acute for the last 15 days
* Patients consenting to participate to the study

Exclusion Criteria for patients of all groups:

* Patients/Healthy volunteers under 18 years old
* Patients/Healthy volunteers protected by the law
* Patients/Healthy volunteers not consenting to participate to the study after information
* Patients with inflammatory pathology or infectious acute intercurrent pathology in the last 15 days before inclusion
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 : Adult with SSc Group 2 : Adult with other connective tissue disease Group 3 : Healthy adult volunteer
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2028-10-27 (Estimated); Study Completion 2029-04-27 (Estimated)

PRIMARY OUTCOMES:
Quantification of Neutrophil Extracellular Traps (NETs) generated after stimulation of neutrophils in vitro by serum from SSC, SLE and healthy controls. | Day 0
  Comparative analysis of the quantity of Neutrophil Extracellular Traps (NETs) generated after stimulation of neutrophils in vitro by serum from SSC, other connective tissue diseases and healthy controls. Neutrophils from SSC, other connective tissue diseases and healthy subjects will be used.

SECONDARY OUTCOMES:
Analysis of the composition of Neutrophil Extracellular Traps (NETs) | Day 0
  Comparative analysis of the composition of Neutrophil Extracellular Traps (NETs) generated after stimulation of neutrophils in vitro by serum from SSC, other connective tissue diseases and healthy controls. Neutrophils from SSC, other connective tissue diseases and healthy subjects will be used.
Analysis of the cytokines influencing Neutrophil Extracellular Traps NETs production in vitro | Day 0
  Comparative analysis of the quantity of Neutrophil Extracellular Traps (NETs) generated after stimulation of neutrophils from SSC patients in vitro by differents cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Didier K, Giusti D, Le Jan S, Terryn C, Muller C, Pham BN, Le Naour R, Antonicelli FD, Servettaz A. Neutrophil Extracellular Traps Generation Relates with Early Stage and Vascular Complications in Systemic Sclerosis. J Clin Med. 2020 Jul 7;9(7):2136. doi: 10.3390/jcm9072136. PMID 32645862